CLINICAL TRIAL: NCT01479504
Title: A Multicenter Trial Evaluating the Efficacy and Safety of Nedaplatin Plus Docetaxel in Neoadjuvant Chemotherapy Followed by Nedaplatin in Concurrent Chemoradiation for Patients With Locoregionally Advanced Nasopharyngeal Carcinoma
Brief Title: A Multicenter Trial Evaluating the Efficacy of Nedaplatin in Patients With Locoregionally Advanced Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangxi Medical University (Other)
Collaborators: People's Hospital of Guangxi Zhuang Autonomous Region (Other); 303rd Hospital of the People's Liberation Army (Other); Nanning Second People's Hospital (Other); Guangxi Traditional Chinese Medical University (Other); Guilin Medical College (Other); Guangxi Naxishan Hospital (Other); Liuzhou Workers' Hospital (Other Government); LiuZhou People's Hospital (Other); Liuzhou Hospital of Traditional Chinese Medicine (Other); Liuzhou Cancer Hospital (Unknown); Liuzhou Railway hospital (Unknown); First People's Hospital of Yulin (Other); The Red Cross hospital of YuLin (Unknown); Guigang People's Hospital (Other); Wuzhou Red Cross Hospital (Other)
Responsible Party: Principal Investigator, Wang Rensheng, Director, Guangxi Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GuangxiMU
Record Dates: First submitted 2011-11-16; First posted 2011-11-24 (Estimated); Last update posted 2011-11-28 (Estimated); Status verified 2011-10

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma; neoadjuvant chemotherapy; concurrent chemoradiotherapy; Nedaplatin
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — nedaplatin; Docetaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1A(nedaplatin and IMRT) (Experimental): neoadjuvant chemotherapy using nedaplatin plus docetaxel followed by concurrent chemotherapy using nedaplatin and Intensity-modulated Radiation Therapy(IMRT)
  Interventions: Drug: nedaplatin and docetaxel
- 1B(cisplatin and IMRT) (Active Comparator): neoadjuvant chemotherapy using cisplatin plus docetaxel followed by concurrent chemotherapy using cisplatin and Intensity-modulated Radiation Therapy(IMRT)
  Interventions: Drug: cisplatin and docetaxel
- 2A(nedaplatin and CRT) (Experimental): neoadjuvant chemotherapy using nedaplatin plus docetaxel followed by concurrent chemotherapy using nedaplatin and conventional fractionation radiotherapy(CRT)
  Interventions: Drug: nedaplatin and docetaxel
- 2B((cisplatin and CRT)) (Active Comparator): neoadjuvant chemotherapy using cisplatin plus docetaxel followed by concurrent chemotherapy using cisplatin and conventional fractionation radiotherapy(CRT)
  Interventions: Drug: cisplatin and docetaxel

INTERVENTIONS:
Drug: nedaplatin and docetaxel — neoadjuvant chemotherapy: nedaplatin 80mg/m2+docetaxel 65 mg/m2/day,every 21 days for 2 cycles before radiotherapy
  concurrent chemotherapy: nedaplatin 40mg/m2,weekly,for 6 cycles during radiotherapy
  Other Names: TN
  Arms: 1A(nedaplatin and IMRT)
Drug: cisplatin and docetaxel — neoadjuvant chemotherapy: cisplatin 80mg/m2+docetaxel 65 mg/m2/day,every 21 days for 2 cycles before radiotherapy
  concurrent chemotherapy: cisplatin 40mg/m2,weekly,for 6 cycles during radiotherapy
  Other Names: TP
  Arms: 1B(cisplatin and IMRT)
Drug: nedaplatin and docetaxel — neoadjuvant chemotherapy: nedaplatin 80mg/m2+docetaxel 65 mg/m2/day,every 21 days for 2 cycles before radiotherapy
  concurrent chemotherapy: nedaplatin 40mg/m2,weekly,for 6 cycles during radiotherapy
  Other Names: TN
  Arms: 2A(nedaplatin and CRT)
Drug: cisplatin and docetaxel — neoadjuvant chemotherapy: cisplatin 80mg/m2+docetaxel 65 mg/m2/day,every 21 days for 2 cycles before radiotherapy
  concurrent chemotherapy: cisplatin 40mg/m2,weekly,for 6 cycles during radiotherapy
  Other Names: TP
  Arms: 2B((cisplatin and CRT))

SUMMARY:
This study is a multicenter trial.The primary objective is to estimate short-term efficacy and acute toxicities of nedaplatin to the combination of docetaxel in neoadjuvant chemotherapy followed by nedaplatin in concurrent chemoradiotherapy, compared to cisplatin to the combination of docetaxel in neoadjuvant chemotherapy followed by cisplatin in concurrent chemoradiotherapy for patients with locoregionally advanced nasopharyngeal carcinoma.

Secondary objectives are to evaluate the overall survival, the distant metastases free survival, and disease free survival of patients with locoregionally advanced nasopharyngeal carcinoma treated with these regimens.Furthermore,analyze the cost-effectiveness of the regimens.

DETAILED DESCRIPTION:
Patients with clinical stage T3-4N1/N2-3 (UICC 7th edition)are divided into two groups according to informed consent:intensity-modulated radiation therapy（IMRT）group and conventional fractionation radiotherapy(CRT)group. Then the patients in IMRT group/CRT group are randomly assigned to receive nedaplatin+docetaxel in neoadjuvant chemotherapy plus nedaplatin alone in concurrent chemoradiotherapy or cisplatin+docetaxel in neoadjuvant chemotherapy plus cisplatin alone in concurrent chemoradiotherapy.Evaluate the overall survival, the distant metastases free survival, and disease free survival of the patients treated with these regimens.Furthermore,analyze the cost-effectiveness of the regimens.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven nasopharyngeal carcinoma for primary treatment with radical intent
* non-keratinizing or undifferentiated type
* clinical stage III-IVb (UICC 7th edition)
* age between 18-70
* satisfactory performance status: Karnofsky scale (KPS) > 70.
* hemoglobin > 100g/L, WBC > 4.0x10*9/L, Plt > 100x10*9/L
* serum creatinine level < 1.6 mg/dL or creatinine clearance ≥ 60 mL/min.
* normal liver function test: Alanine Aminotransferase (ALT)、Aspartate Aminotransferase (AST) <1.5×upper limit of normal (ULN) concomitant with alkaline phosphatase (ALP) ≤2.5×ULN, and bilirubin ≤1.5ULN
* patients must be informed of the investigational nature of this study and give written informed consent.
* anticipated life span more than 6 month

Exclusion Criteria:

* primary treatment with palliative intent
* WHO Type keratinizing squamous cell carcinoma or basaloid squamous cell carcinoma Evidence of distant metastases
* pregnancy or lactation
* history of previous radiotherapy (except for non-melanomatous skin cancers outside intended RT treatment volume).
* prior chemotherapy or surgery (except diagnostic) to primary tumor or nodes
* prior malignancy except adequately treated basal cell or squamous cell skin cancer, in-situ cervical cancer or other cancer for which the patient has been disease-free for 5 years
* any severe intercurrent disease, which may bring unacceptable risk or affect the compliance of the trial, for example, unstable cardiac disease requiring treatment, renal disease, chronic hepatitis, diabetes with poor control (fasting plasma glucose >1.5×ULN), and emotional disturbance.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
complete response (CR) rate | 3 months
  3 months after treatment

SECONDARY OUTCOMES:
Acute toxicities | 2 years
  Acute toxicity will be measured by CTCAE3.0
Overall Survival | 1,3,5 years
  1 years，3 years and 5 years overall survival,disease free survival,distant metastases free survival
cost-effectiveness ratio | 3 months
  Calculate the cost(C) and complete response rate(E) of each group 3 months after treatment,then calculate cost-effectiveness ratio(C/E).

CONTACTS AND LOCATIONS:
Overall Officials: Wang R. sheng, M.D., Study Chair — Department of Radiotherapy，the First Affiliated Hospital of Guangxi Medical University; Wang R sheng, M.D., Principal Investigator — Department of Radiotherapy，the First Affiliated Hospital of Guangxi Medical University; Wu Fang, M.D., Principal Investigator — Department of Radiotherapy，the First Affiliated Hospital of Guangxi Medical University
Locations (1):
- Department of Radiotherapy，the First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi, China